CLINICAL TRIAL: NCT06276244
Title: Trial Readiness and Endpoint Assessment in Congenital and Childhood Myotonic Dystrophy
Acronym: GUP19002
Status: Completed | Type: Observational
Sponsor: Fondazione Serena Onlus - Centro Clinico NeMO Milano (Other)
Collaborators: Bambino Gesù Hospital and Research Institute (Other); Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other); IRCCS Istituto delle Scienze Neurologiche di Bologna (Other); IRCCS Fondazione Stella Maris (Other); Fondazione Mondino (Other); A.O.U. Città della Salute e della Scienza (Other); Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other); Istituto Giannina Gaslini (Other)
Responsible Party: Sponsor
Other Study IDs: NM040-GUP19002
Record Dates: First submitted 2024-01-15; First posted 2024-02-23 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: CDM; ChDM
Keywords: congenital myotonic dystrophy; childhood myotonic dystrophy
MeSH Terms: conditions — Myotonic Dystrophy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — PAX-gene
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Congenital Myotonic Dystrophy (CDM): CDM group:
  1. Age 0-17 years, 11 months of age
  2. A diagnosis of CDM, which is defined as children having symptoms of myotonic dystrophy in the newborn period (<30 days), such as hypotonia, feeding or respiratory difficulty, requiring hospitalization to a ward or to the neonatal intensive care unit for more than 72 hours; and a genetic test confirming an expanded trinucleotide (CTG) repeat in the DMPK gene in the child or mother. An expanded CTG repeat size in the child is considered greater than 200 repeats or E1-E4 classification (E1= 200-500, E2=500-1,000, E3=1,000-1,500, E4>1,500).
- Childhood Muscular Dystrophy (ChDM): ChDM group:
  1. Age 0-17 years, 11 months of age
  2. A diagnosis of ChDM, which is defined as children having symptoms of myotonic dystrophy after day 30 from birth. These may include any delay in psychomotor development, attention deficit disorder, behavioral abnormalities within the spectrum of autistic spectrum disorders, gastrointestinal dysfunction such as persistent constipation or diarrhea and gastroesophageal reflux; and a genetic test confirming an expanded trinucleotide (CTG) repeat in the DMPK gene in the child or mother. An expanded CTG repeat size in the child is considered greater than 200 repeats.

SUMMARY:
Children with congenital myotonic dystrophy (CDM) present at birth with respiratory insufficiency, talipes equinovarus, feeding difficulties and hypotonia. There is a 30% mortality rate in the first year of life. Children with childhood onset myotonic dystrophy present with symptoms later on but soon develop behavioural difficulties and learning difficulties and are at risk for autistic features and gastrointestinal symptoms. The ability to conduct a therapeutic trial in children with CDM or ChDM is directly limited by the lack of available data regarding appropriate clinical endpoints and biomarkers. Whereas there is an active Italian collaboration recruiting adults with DM1 to study muscle and multisystem aspects in this population, there is no active network in Italy involved in the pediatric population with DM1. Though the underlying mechanism is the same in adult DM1, in CDM and ChDM there are specific challenges to the pediatric population. The aim of this project is to coordinate the Italian Child Neurologist actively involved with CDM and ChDM in a common effort of standardizing protocols and procedures to be applied in the care of these patients. Specific aims are to collect functional measures and clinical information over time to define clinically meaningful endpoints and outcome measures in preparation for international therapeutic clinical trials. This project will contribute to the ongoing international study in CDM by recruiting additional patients from all over Italy and will extend the investigations to the childhood onset forms as an additional add-on pilot study in view of potential treatment options. The investigators expect that the Italian network, with Telethon support, will provide the necessary backbone for trial readiness in the pediatric population both at the national and international levels.

DETAILED DESCRIPTION:
observational prospective study

ELIGIBILITY:
Inclusion criteria, CDM group:

1. Age 0-17 years, 11 months of age
2. A diagnosis of CDM, which is defined as children having symptoms of myotonic dystrophy in the newborn period (<30 days), such as hypotonia, feeding or respiratory difficulty, requiring hospitalization to a ward or to the neonatal intensive care unit for more than 72 hours; and a genetic test confirming an expanded trinucleotide (CTG) repeat in the DMPK gene in the child or mother. An expanded CTG repeat size in the child is considered greater than 200 repeats or E1-E4 classification (E1= 200-500, E2=500-1,000, E3=1,000-1,500, E4>1,500).

Inclusion criteria, ChDM group:

1. Age 0-17 years, 11 months of age
2. A diagnosis of ChDM, which is defined as children having symptoms of myotonic dystrophy after day 30 from birth. These may include any delay in psychomotor development, attention deficit disorder, behavioral abnormalities within the spectrum of autistic spectrum disorders, gastrointestinal dysfunction such as persistent constipation or diarrhea and gastroesophageal reflux; and a genetic test confirming an expanded trinucleotide (CTG) repeat in the DMPK gene in the child or mother. An expanded CTG repeat size in the child is considered greater than 200 repeats.

Exclusion criteria, CDM and ChDM groups:

1. Any other non-DM1 illness that would interfere with the ability or results of the study in the opinion of the site investigator
2. Significant trauma within one month
3. Internal metal or devices (exclusion for DEXA component)
4. Unable to walk more than 50 feet if over the age of 3.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Please refer to the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2020-07-08 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Physical function | From Baseline (T0) to Days 1080
  Measures of right grip strength using hand-held myometry
Physical function | From Baseline (T0) to Days 1080
  Oral facial strength as measured by lip-force meter
Cognitive-behavioral and Quality of Life | From Baseline (T0) to Days 1080
  Total score and subscores from the CCMDHI
Cognitive-behavioral and Quality of Life | From Baseline (T0) to Days 1080
  BRIEF total scores
Biomarkers | From Baseline (T0) to Days 1080
  Muscle RNA splicing changes
Biomarkers | From Baseline (T0) to Days 1080
  Lean muscle mass

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Serena Onlus - Centro Clinico NeMO Milano, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided